CLINICAL TRIAL: NCT02759484
Title: MATCH2: The Multi-clinic Action Trial to Control Hyperglycemia and Hypertension
Brief Title: Multi-clinic Action Trial to Control Hyperglycemia and Hypertension
Acronym: MATCH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12052906
Record Dates: First submitted 2015-12-18; First posted 2016-05-03 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: CHWs; Health Education; Disease Self Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home Based Enhanced Education (Experimental): The Home Based Enhanced Education arm consists of a diabetes self-management curriculum delivered by Community Health Workers in the participant's home.
  Interventions: Behavioral: Home Based Enhanced Education
- Clinic Based Enhanced Education (Active Comparator): The Clinic Based Enhanced Education arm consists of group diabetes self-management education, delivered by a Certified Diabetes Educator, plus mailed diabetes self-management education.
  Interventions: Behavioral: Clinic Based Enhanced Education

INTERVENTIONS:
Behavioral: Home Based Enhanced Education — The Home Based Enhanced Education arm consists of a diabetes self-management curriculum delivered by Community Health Workers in the participant's home. Participants receive 24 visits: 12 biweekly visits in the first 6 months, followed by 12 monthly visits in months 6 through 18 of the study. The self-management program is derived from two pragmatic evidence-based frameworks for behavioral change.
  Other Names: Community Health Worker intervention (CHW)
  Arms: Home Based Enhanced Education
Behavioral: Clinic Based Enhanced Education — The Clinic Based Enhanced Education arm consists of two two-hour-long sessions of group diabetes self-management education, delivered by a Certified Diabetes Educator. Participants in this arm will also receive 24 newsletters with diabetes self-management education.
  Other Names: Diabetes Educator intervention
  Arms: Clinic Based Enhanced Education

SUMMARY:
The MATCH2 Study (The Multi-clinic Action Trial to Control Hyperglycemia and Hypertension) is a randomized controlled trial comparing two educational approaches to improve glucose and blood pressure control in African American and Latino adults with type 2 diabetes. The study is being designed and implemented using a Community Based Participatory Research approach to optimize the two educational approaches. One approach, Enhanced Home Based Education, adapts a Community Health Worker (CHW) intervention from the protocol of the prior Mexican-American Trial of Community Health workers (MATCH). The other approach, Enhanced Clinic Based Education, uses a Certified Diabetes Educator (CDE) to deliver dietary and general self-management education. The study seeks to determine if Community Health Workers working as part of the primary care clinical team can reduce health disparities and improve outcomes among patients with type 2 diabetes.

DETAILED DESCRIPTION:
MATCH2, a randomized controlled trial, will test if the optimized CHW-delivered intervention can reduce both Hemoglobin A1c levels and blood pressure at eighteen months in persons with uncontrolled diabetes, as compared to a CDE-delivered group educational program. Follow-up six months after the completion of the intervention will evaluate the sustainability of any gains. MATCH2 will use precise measures of diet (food frequency questionnaires) and physical activity (accelerometry) to identify intermediate behaviors and processes that mediate significant improvements in glycemic and blood pressure control.

Patients/participants will be recruited from three participating urban primary care safety net clinics to join MATCH2 if patients meet the inclusion and exclusion conditions (see criteria section below). Eligible patients interested in participation will have a baseline visit scheduled. Baseline assessments may be conducted either at the clinic, the participant's home, or the Rush Prevention Center, at the patient's preference. At the baseline visit, the research assistant will obtain informed consent for the study as approved by the Institutional Review Boards (IRB) of participating institutions. The baseline assessment will include the following measures: demographics, clinical data, glycemic control, blood pressure, total caloric and sodium intake, physical activity, medication adherence, clinic attendance, quality of life, patient activation, depression and social support.

A randomization scheme based on permuted randomized blocks of size 4 and 6 will be used, stratified by clinic. Randomization schedules will be developed by the study Biostatistician and the Data Management Team will assign participants to treatment or control groups accordingly.Of the investigative team, the Principal Investigator, identified Key Co-Investigators and all research assistants will be blinded to the patient's group assignment while remaining research team: the Community Health Workers (blinded to study hypothesis), selected Key Co-Investigators, Site Principal Investigators, and Data Management Team will be unblinded.

Participants will know the study condition to which participants have been assigned. As with the CHW interventionists, participants will be blinded to the study hypothesis. Consent and recruitment forms will all state that "The MATCH2 trial is comparing two clinic-based approaches to improve control of high blood sugar and high blood pressure in people with type 2 diabetes. Some evidence suggests that approaches such as health classes led by a diabetes educator, coaching by Community Health Workers, and printed diabetes education materials may help improve outcomes for people with uncontrolled diabetes.

ENHANCED HOME-BASED EDUCATION CONDITION: CHW Interventionists deliver diabetes self-management curriculum in the participant's home or other preferred setting.

MATCH2 Trained CHW Interventionists will work closely with patients to deliver a participant-centered intervention derived from two pragmatic evidence-based frameworks for behavioral change [Motivational Interviewing (MI) and Kate Lorig's Chronic Disease Self-Management approach]. 24 total in-person visits will be conducted; six primary topics will be covered multiple times over an 18-month period. No more than two topics will be addressed at any visit. The sequence in which topics are delivered is determined by participant need, preference, and interest. The six primary topics are:

1. Check glucose daily and know the goal.
2. Check blood pressure daily and know the goal.
3. Understand medications and take medications as prescribed.
4. Engage in 30 minutes of physical activity every day.
5. Enjoy a healthy natural diet with vegetables, fruit, and fiber.
6. Communicate any concerns to the health care team.

At each visit, CHWs will help participants develop a self-management Action Plan around one of the six topics, and support problem solving behaviors to address barriers to completing the Action Plan. Behavioral self-management skills will be taught by the CHW and practiced with the participant at each visit. CHWs will monitor the clinic attendance of participants and will advise and assist participants with making appointments with their primary care providers at least once every 4 months. CHWs will also play an active role in communicating the progress of their participants to the primary care providers using the clinic Electronic Medical Record.

ENHANCED CLINIC-BASED EDUCATION CONDITION: Participants will receive group diabetes self-management education, consistent with current Medicare guidelines for diabetes education. A Certified Diabetes Educator will deliver the two class sessions (each two hours) covering basic topics: diabetes (including self-management) and nutrition. Participants will also receive 24 bilingual educational newsletters: twelve during the first six months and then once a month between 6 and 18 months. The newsletters, called "Diabetes Action", cover the same six self-management topics listed previously.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus with A1c greater than or equal to 7.0
* At least 18 years of age and capable of giving informed consent in either English or Spanish
* Primary care received through a participating clinic
* Participants must identify themselves as either Black / African American race or Hispanic / Latino ethnicity

Exclusion Criteria:

* Have end-stage renal disease, stroke, or other major end-organ complication of diabetes
* Require chronic prednisone or other systemic corticosteroid use
* Are receiving treatment for a major psychiatric disorder (i.e. schizophrenia)
* Live in a household with someone who is already a randomized study participant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2015-03; Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Glycemic Control | Up to 18 months post randomization
  Glycemic control will be determined by Hemoglobin A1c, measured on a fingerstick collected Dried Blood Spot test, and analyzed by an independent reference lab.
Blood Pressure Control | Up to 18 months post randomization
  Blood Pressure (BP) will be measured three times using an automated blood pressure cuff with the participant in a seated position. Mean Arterial Pressure will be calculated by the standard formula: Diastolic BP + 1/3 (Systolic BP - Diastolic BP)] .

SECONDARY OUTCOMES:
Maintenance of Glycemic Control | Up to 24 months post randomization
  Glycemic control will be determined by Hemoglobin A1c, measured on a fingerstick collected Dried Blood Spot test, and analyzed by an independent reference lab.
Maintenance of Blood Pressure Control | Up to 24 months post randomization
  Blood Pressure (BP) will be measured three times using an automated blood pressure cuff with the participant in a seated position. Mean Arterial Pressure will be calculated by the standard formula: Diastolic BP + 1/3 (Systolic BP - Diastolic BP)] .
Intermediate Behavior: Dietary Adherence | Up to 18 months
  Repeated 24-hour dietary recalls using the Nutrition Data System for Research (NDSR)
Intermediate Behavior: Physical Activity | Up to 18 months
  Accelerometer, worn for one week.
Intermediate Behavior: Medication Adherence | Up to 18 months
  Morisky 8-item questionnaire (MMAS-8)

OTHER OUTCOMES:
Intervention Costs | Up to 24 months
  Participant and system costs will be collected including, but not limited to: all intervention costs, participant time and travel, clinic visits, emergency department encounters, hospitalizations, and medication costs.

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Rothschild, MD, Principal Investigator — Rush University Medical Center
Locations (3):
- United States (3):
  - Rush University Internists, Chicago, Illinois
  - Erie Family Health Center, Chicago, Illinois
  - Cicero Health Center of Cook County, Cicero, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data from the trial will be made available to qualified investigators following completion of the trial and all major data analyses.